CLINICAL TRIAL: NCT01165892
Title: Pulmonary MR Angiography and Lower Extremity MR Venous Imaging Using a Single Dose of Gadofosveset (Ablavar)
Brief Title: Pulmonary MR Angiography and Lower Extremity MR Venous Imaging Using Gadofosveset (Ablavar)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-0567
Record Dates: First submitted 2010-07-02; First posted 2010-07-20 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; contrast agent
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gadofosveset Triodium — Use of 0.03 mmol/Kg of gadofosveset trisodium (Ablavar)once with intravascular half life of up to 1 hr and optimal arterial imaging out to 20-30 minutes.
  Other Names: Ablavar

SUMMARY:
The use of the contrast agent, Ablavar, will help with the diagnosis of pulmonary embolism in magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Specific Aim 1: To assess first-pass SNR and CNR of pulmonary MR angiography performed with 0.03 mmol/Kg of intravenous gadofosveset trisodium.

Hypothesis: Use of 0.03 mmol/Kg of gadofosveset trisodium in gradient recalled echo pulmonary MR angiography will provide a pulmonary artery SNR and CNR equal to or better than the SNR and CNR obtained using the same MR technique with 0.2 mmol/Kg of a conventional contrast agent (gadopentetate dimeglumine) and equal to or better than 0.1 mmol/Kg of intravenous gadobenate dimeglumine. Data will be compared to SNR and CNR of pulmonary MR angiogram images obtained at Washington University as part of the PIOPED III study.

Specific Aim 2: To assess SNR and CNR of breath-hold pulmonary MR imaging obtained immediately after the original first-pass breath-hold pulmonary MR angiography.

Hypothesis: SNR and CNR of pulmonary MR angiography performed immediately after first-pass breath-hold pulmonary MR angiography will be at least equal to the SNR and CNR obtained using the same MR technique with 0.2 mmol/Kg of a conventional contrast agent (gadopentetate dimeglumine) and at least equal to 0.1 mmol/Kg of intravenous gadobenate dimeglumine.

Specific Aim 3: To assess SNR and CNR of lower extremity MR venogram (MRV) performed immediately after the two pulmonary MR angiograms, described above.

Hypothesis: SNR and CNR of passive lower extremity MRV performed after pulmonary MR angiography will be equal to or better than the SNR and CNR obtained using the same passive MRV technique with 0.2 mmol/Kg of a conventional contrast agent or 0.1 mmol/Kg of gadobenate dimeglumine. Again, data will be compared to SNR and CNR of lower extremity

ELIGIBILITY:
Inclusion Criteria:

1. Patient that have pulmonary embolism.
2. 18 yrs of age and older

Exclusion Criteria:

1. allergy to gadolinium based contrast.
2. allergy to iodated based contrast.
3. renal insufficiency (GFR < 60 mL/min?1.73m2)
4. pregnant or nursing
5. contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Imaging Outcome | Upon imaging
  Assessment of imaging parameters such as SNR, CNR

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Woodard, M.D., Principal Investigator — Washington University School of Medicine